CLINICAL TRIAL: NCT02542995
Title: Creating Healthy Workplaces: Improving Outcomes for Providers and Patients
Brief Title: Creating Healthy Work Places (HWP) Study
Acronym: HWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); University of Wisconsin, Madison (Other); Marshfield Clinic Research Foundation (Other); New York University (Other); Loyola University School of Medicine (Unknown); University of Alabama, Tuscaloosa (Other); University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Mark Linzer, Division Director of General Internal Medicine, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AHRQ 1R18-HSO18160-03
Record Dates: First submitted 2015-08-27; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-intervention (No Intervention): Usual clinical conditions
- Intevention (Other): QI interventions and got to see their own survey data - examples include:
  Workflow redesign:
  Medical Assistant (MA) data entry Improved clinic efficiency projects Assessed workflow with staff Provided time for MAs and RNs to perform tasks Paired MAs and providers Non-physician staff assist with forms
  Communication improvement:
  Improved teamwork Improved communication between provider groups Routine clinician meetings discussing meaningful topics Survey of providers for "wish list" of issues Routine emails from leaders Clinicians meeting with leaders
  Chronic disease QI projects:
  Establishing quality metrics with clinician input Automated Rx refill line Med reconciliation project Screening project for diabetics Screening for depression Improved patient portals
  Interventions: Other: QI interventions

INTERVENTIONS:
Other: QI interventions — Intervention categories: communication improvement, chronic disease QI projects (for patients), workflow redesign
  Arms: Intevention

SUMMARY:
The health of the public depends upon smoothly functioning physician offices that promote the health of both workers and their patients. This study targets ambulatory health care offices with rapid paced, chaotic environments. Investigators will measure adverse outcomes for providers and staff (e.g., stress and burnout), the impact these have on quality of care for hypertensive, diabetic and depressed patients, and identify areas where practice redesign to create "healthy workplaces" improves these outcomes.

DETAILED DESCRIPTION:
The context in which primary care is delivered is rarely evaluated as part of quality improvement initiatives or research projects. Data from the MEMO Study (Minimizing Error, Maximizing Outcome) confirm a relationship between the work environment, provider reactions, and patient care. Time pressure is associated with physician satisfaction, stress, burnout, and intent to leave as well as lower quality care for hypertensive patients. Lack of values alignment between physicians and leaders is associated with physician satisfaction, stress, burnout, and intent to leave as well as poorer diabetes care and fewer prevention activities. Thus, providers are not the only ones at risk in adverse work conditions. An important coexisting factor is the impending primary care physician shortage. Less than optimal work conditions are associated with physician intent to leave and with reduced medical student interest in primary care. This randomized study assessed the impact of applying a novel quality improvement strategy designed to create "healthy workplaces".

The investigators hypothesized that addressing adverse primary care work conditions (workflow, work control, organizational culture) would lead to greater clinician participation in programs to improve health care delivery. As part of MEMO, the investigators developed the Office and Work Life (OWL) measurement tool. The OWL assesses the primary care workplace and identifies specific working conditions that impact provider outcomes and quality of care. The current proposal assessed the ability of the OWL and a focused QI process to facilitate changes in the work environment and improve outcomes for providers and patients.

Thirty-four primary care clinics were recruited in New York City and the upper Midwest. Physicians, physician assistants, and nurse practitioners (n=165) were surveyed to collect OWL data on provider outcomes, and organizational structure and culture. Managers were asked to provide information on clinic structure, policies and procedures. Eight patients per provider (n=1131) with hypertension and /or diabetes will be surveyed on health literacy, quality of life, medication compliance, satisfaction, and trust. Patient charts were audited to assess hypertension and diabetes management. The data was then compiled into an OWL measure for each clinic.

34 clinics were randomized. Local leaders, providers, and staff in 17 intervention clinics received their OWL measure and discussed the successes and challenges to care illustrated by the data. Assisted by the study team, they developed QI plans focusing on workplace variables that investigators found contributed to care quality: time pressure, work control, work pace (chaos), and organizational culture. Twelve months later (Aug. 2012 - Jan. 2013), OWL data was recollected in all 34 clinics and compared.

New OWL data was fed back to personnel in the 17 intervention clinics to formalize its role in continuous QI processes. Control clinics received their OWL data at study end. Subsets of data were analyzed to determine the best ways to modify the work environment to improve outcomes for underrepresented groups (women and minority providers and minority patients).

ELIGIBILITY:
Inclusion Criteria:

* 18+,
* have a primary care provider at one of enrolling institutions,
* have a primary care visit within year of enrollment

Exclusion Criteria:

* Deceased,
* inability to communicate (hard of hearing), etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1296 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Medical provider stress and burnout | Provider outcomes were measured approximately one year after the interventions
  Survey tools: to measure provider stress and burnout developed (for providers), the survey tools were used in the MEMO study and have 1-5 scales.
Patient satisfaction with care | Patient satisfaction was measured at baseline and approxmiaetly one year after the interventions
  Survey tool (patients self reported), the survey tools were used in the MEMO study and have 1-5 scales.
Patient quality of care | Patient quality of care was measured at baseline and approxmiaetly one yr after the interventions
  Chart audits

SECONDARY OUTCOMES:
Provider turnover (cost) | Provider turnover (cost) was mesasured about one year after the interventions
  Clinic managers were given a survey (similar to the ones used by provider and patients) and asked to document the clinic staff make up, how often positions were posted and the length of time of the posting to help assess cost of provider turnover.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Linzer, MD, Principal Investigator — MMRF

REFERENCES:
- [Derived] Khullar D, Prasad K, Neprash H, Poplau S, Brown RL, Williams ES, Audi C, Linzer M. Factors associated with patient trust in their clinicians: Results from the Healthy Work Place Study. Health Care Manage Rev. 2022 Oct-Dec 01;47(4):289-296. doi: 10.1097/HMR.0000000000000336. Epub 2022 Feb 17. PMID 35170482
- [Derived] Linzer M, Poplau S, Brown R, Grossman E, Varkey A, Yale S, Williams ES, Hicks L, Wallock J, Kohnhorst D, Barbouche M. Do Work Condition Interventions Affect Quality and Errors in Primary Care? Results from the Healthy Work Place Study. J Gen Intern Med. 2017 Jan;32(1):56-61. doi: 10.1007/s11606-016-3856-2. Epub 2016 Sep 9. PMID 27612486